CLINICAL TRIAL: NCT00000345
Title: Evaluation of Lofexidine for Treatment of Opiate Withdrawal
Brief Title: Evaluation of Lofexidine for Treatment of Opiate Withdrawal - 10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NIDA-3-0010-10; Y01-3-0010-10
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1997-09

CONDITIONS: Opioid-Related Disorders
Keywords: opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine

INTERVENTIONS:
Drug: Lofexidine

SUMMARY:
The purpose of this study is to assess the safety of lofexidine in the treatment of opiate-dependent individuals.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Meet DSM-IV criteria for opiate dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nuring women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical condtions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-04

PRIMARY OUTCOMES:
Opiate withdrawal
Adverse effect measures
Craving of opiates
Liking of opiates
Efficacy of lofexidine
Euphoria

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States